CLINICAL TRIAL: NCT04020939
Title: The Role of Indocyanine Green Angiography Fluorescence on Intestinal Resections in Pediatric Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Nelson Piche, Pediatric Surgeon, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-2359
Record Dates: First submitted 2019-07-02; First posted 2019-07-16 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Intestinal Atresia; Necrotizing Enterocolitis; Hirschsprung Disease; Gastroschisis; Intestinal Obstruction; Incarcerated Hernia; Intussusception; Malrotation; Volvulus; Meconium Ileus; Intestinal Perforation; Trauma
Keywords: SPY imaging; indocyanine green; pediatric surgery; ICG; intestinal resections; intestinal perfusion
MeSH Terms: conditions — Intestinal Atresia; Enterocolitis, Necrotizing; Hirschsprung Disease; Gastroschisis; Intestinal Obstruction; Intussusception; Volvulus Of Midgut; Intestinal Volvulus; Meconium Ileus; Intestinal Perforation; Wounds and Injuries | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing intestinal resections (Experimental): * Interventions to be administered: indocyanine green intravenous injection and subsequent visualisation of intestinal viability under fluorescence
  * Drug:
  Indocyanine green dye (ICG) Dosage: 0.5 mg/kg (diluted with aqueous solution) Maximum: 2 mg/kg Frequency: maximum of 3 boluses Duration: intraoperative use only
  Interventions: Device: SPY imaging; Drug: Indocyanine Green

INTERVENTIONS:
Device: SPY imaging — Use of the SPY Pinpoint imaging device to evaluate intraoperative intestinal perfusion in children.
  Other Names: SPY PinPoint
Drug: Indocyanine Green — Intravenous injection of indocyanine green to evaluate the intestinal perfusion.
  Other Names: ICG; IC-Green

SUMMARY:
Background: Intestinal resections are commonly performed in the pediatric population. Perfusion of the bowel is one of the most important factors determining the viability of an intestinal anastomosis. Up to date, no ideal method to assess intestinal perfusion has proven its superiority.

Objectives:

Primary: The aim of this study is to establish the feasibility and impact of the use of indocyanine green technology on intestinal resection margins during elective and emergency pediatric surgeries.

Secondary: The secondary outcomes of interest include collection of adverse events and difficulties encountered with the use of the indocyanine green (ICG) technology. Postoperative surgical complications will also be recorded.

Study Design: An open observational clinical study will be performed by using a clinical drug (indocyanine green) and medical device (SPY Fluorescence Imaging) to assess intraoperatively intestinal perfusion in a specific pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 16 years old
* Admitted between September 2019 and September 2020
* Patients undergoing a surgery at CHUSJ
* Any diagnosis requiring intra-abdominal intestinal resection (including stoma reversal)
* Written informed consent form from the parents or legal guardian

Exclusion Criteria:

* Patients > 16 years old
* Patients with known allergy or sensitivity to iodine
* Patients with known kidney or liver failure
* Patients with known severe cardiac or pulmonary diseases
* Informed consent unobtained or impossible due to refusal of parents, language barrier, or diminished comprehension

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
SPY System utility in intestinal resections in Pediatric Surgery | 1 year
  To demonstrate the utility of intra-operative evaluation of intestinal viability using the SPY Fluorescence Imaging System to optimize the location of the resection margins in pediatric surgeries necessitating intestinal resections.
  - Rate of intestinal resection margins modifications by using the SPY technology

SECONDARY OUTCOMES:
Surgical complications | 1 year
  * Number of anastomotic leaks
  * Number of strictures
  * Number of bowel obstructions
Length of stay | 1 year
  In days
Operative time | 30 days
  In minutes
Estimated blood losses | 30 days
  In ml
Need for additional reoperations | 1 year
  Number
Need for additional radiology interventions | 1 year
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Piché, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No